CLINICAL TRIAL: NCT02900833
Title: Neutrophil Activation in Acute Ischemic Stroke Patients Treated With Endovascular Therapy
Brief Title: Impact of Neutrophil Activation in Acute Ischemic Stroke Patients Treated With Endovascular Therapy
Acronym: NEUTROSTROKE
Status: Active, not recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JDS_2015_46
Record Dates: First submitted 2016-09-07; First posted 2016-09-14 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical and experimental data suggest that neutrophil activation and extravasation are deleterious in acute ischemic stroke (AIS) involving an increased risk of unfavorable outcome and hemorrhagic transformation (HT). However, clinical trials targeting neutrophil recruitment in AIS patients were negative. Recently, an experimental study has shown that neutrophil activation and transmigration begin immediately after the occlusion. Inhibition of neutrophil recruitment several hours after the start of ischemia appears therefore too late to have a clinical relevance.

The objective is to study the time dependent impact of neutrophils in AIS and the predominant mediators in each time point to identify the appropriate therapeutic target and time window.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years old
* acute ischemic stroke secondary to a large vessel occlusion.
* Patients hospitalized for endovascular therapy.

Exclusion Criteria:

* Pregnant or breast feeding patient
* patient under legal protection
* Patient opposition to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke secondary to a large vessel occlusion, undergoing endovascular therapy.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
neutrophil counts | before recanalization
  Plasma neutrophil activation bio-markers
neutrophil counts | immediately after recanalization
  Plasma neutrophil activation bio-markers
neutrophil counts | 24 hours after recanalization
  Plasma neutrophil activation bio-markers
neutrophil protease counts | before recanalization
recanalization score | immediately after endovascular procedure
  Thrombolysis in Cerebral Infarction classification (TICI)
acute ischemic stroke etiology | within 24 hours after endovascular procedure
  as defined by the Trial of Danaparoid (ORG10172) in Acute Stroke Treatment (TOAST classification)
severity of neurologic symptoms | baseline
  National Institutes of Health Stroke Scale (NIHSS)
disruption of the blood-brain-barrier | within 24 hours after endovascular procedure
  diagnosis on cerebral Computerized Tomography
brain haemorrhage | 24 hours after endovascular procedure
  National Institutes of Health Stroke Scale (NIHSS)
Recovery of motor function after stroke | 3 months
  modified Rankin scale
mortality | 3 months
adhesion molecules counts | before recanalization
adhesion molecules counts | immediately after recanalization
adhesion molecules counts | 24 hours after recanalization
free plasma DNA counts | before recanalization
free plasma DNA counts | immediately after recanalization
free plasma DNA counts | 24 hours after recanalization
neutrophil protease counts | immediately after recanalization
neutrophil protease counts | 24 hours after recanalization

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe DESILLES, MD, Principal Investigator — Fondation OPH A de Rothschild; Mikael MAZIGHI, MD, PhD, Study Chair — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France

REFERENCES:
- [Derived] Boutelier A, Ollivier V, Mazighi M, Kyheng M, Labreuche J, Brikci-Nigassa N, Solo Nomenjanahary M, Delvoye F, Maier B, Paquet C, Ho-Tin-Noe B, Desilles JP. Acute astrocytic reaction is associated with 3-month functional outcome after stroke treated with endovascular therapy. Eur Stroke J. 2024 Dec;9(4):952-958. doi: 10.1177/23969873241256813. Epub 2024 Jun 6. PMID 38845167